CLINICAL TRIAL: NCT05855590
Title: Efficacy of Tranexamic Acid in Debridement Surgery of Burns on the Volume of Bleeding in Transfusion Requirements at Centro Medico de Occidente'
Brief Title: Tranexamic Acid in Debridement Surgery of Burns on the Volume of Bleeding in Transfusion Requirements
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Tranexamic project
Record Dates: First submitted 2023-03-30; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Burns
Keywords: burns
MeSH Terms: conditions — Burns | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, prospective trial to establish the effect of intraoperative tranexamic acid in early surgical debridement of severe burns. The study was carried out between the months of January 2022 to December 2022.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tranexamic acid (Experimental): A total of 20 patients were included: 9 patients in the tranexamic acid group
  Interventions: Drug: Tranexamic acid
- placebo (Placebo Comparator): A total of 20 patients were included: 11 patients in the control group using 0.9% isotonic saline solution.
  Interventions: Other: 0.9% isotonic saline solution

INTERVENTIONS:
Drug: Tranexamic acid — 10mg/kg intravenous single dose
  Arms: tranexamic acid
Other: 0.9% isotonic saline solution — 100 ml intravenous single dose
  Arms: placebo

SUMMARY:
Tranexamic acid in debridement surgery of burns on the volume of bleeding in transfusion requirements

DETAILED DESCRIPTION:
A randomized, double-blind, prospective trial was conducted to establish the effect of intraoperative tranexamic acid in the early surgical debridement of severe burns. The study was carried out between the months of January 2022 and December 2023.

ELIGIBILITY:
Inclusion Criteria:

1. First-time patients undergo surgical debridement of their burns.
2. A burn percentage of 10-30% of burned body surface area
3. Patients over 18 years of age
4. Patients under 40
5. IMSS beneficiaries

Exclusion Criteria:

1. Burned patients with previous surgical debridement.
2. Patients with co-morbids.
3. Patients with a history of drug hypersensitivity.
4. Patients with kidney disease.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Compare the group with tranexamic acid with the group with saline solution. | The time frame: the total time of the study is during the first day, only one dose will be given, and they will be compared at 24 hours.
  The differences between the groups at the beginning of the study were evaluated with the Student's t test for continuous variables, and the proportions were compared with the Chi2 or Fisher test.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Médico Nacional de Occidente, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dominguez A, Alsina E, Landin L, Garcia-Miguel JF, Casado C, Gilsanz F. Transfusion requirements in burn patients undergoing primary wound excision: effect of tranexamic acid. Minerva Anestesiol. 2017 Apr;83(4):353-360. doi: 10.23736/S0375-9393.16.10992-7. Epub 2016 Nov 9. PMID 27827518
- [Background] K S A, Kumar P, Subair M, Sharma RK. Effect of single dose intravenous tranexamic acid on blood loss in tangential excision of burn wounds - A double blind randomised controlled trial. Burns. 2022 Sep;48(6):1311-1318. doi: 10.1016/j.burns.2021.08.021. Epub 2021 Aug 30. PMID 34952736
- [Background] Brown NJ, Choi EH, Gendreau JL, Ong V, Himstead A, Lien BV, Shahrestani S, Ransom SC, Tran K, Tafreshi AR, Sahyouni R, Chan A, Oh MY. Association of tranexamic acid with decreased blood loss in patients undergoing laminectomy and fusion with posterior instrumentation: a systematic review and meta-analysis. J Neurosurg Spine. 2021 Nov 5;36(4):686-693. doi: 10.3171/2021.7.SPINE202217. Print 2022 Apr 1. PMID 34740174
- [Result] Tapking C, Hundeshagen G, Kirchner M, Fischer S, Kneser U, Bliesener B. Tranexamic acid reduced blood transfusions in acute burn surgery: A retrospective case-controlled trial. Burns. 2022 May;48(3):522-528. doi: 10.1016/j.burns.2022.03.002. Epub 2022 Mar 16. PMID 35339324